CLINICAL TRIAL: NCT03210610
Title: Measurement of Colchicine Levels in the Serum of FMF Patients
Brief Title: Colchicine Levels in the Serum of FMF (Familial Mediterranean Fever) Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Merav Lidar, Director, Head of rheumatology clinic, Principal Investigator, Clinical Professor, Sheba Medical Center
Other Study IDs: 3997-17-SMC
Record Dates: First submitted 2017-06-29; First posted 2017-07-07 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: FMF; Colchicine Resistance; Colchicine Toxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FMF patients: fmf patients under a constant colchicine dose
  Interventions: Diagnostic Test: colchicine level measurement

INTERVENTIONS:
Diagnostic Test: colchicine level measurement — levels of colchicine will be measured in FMF patients taking colchicine

SUMMARY:
in this study the investigators will measure the colchicine trough levels in 80 FMF patients taking stable doses of colchicine

DETAILED DESCRIPTION:
80 FMF patients will enroll: 20 taking 1 mg colchicine a day 20 taking 1.5 mg colchicine a day 20 taking 2 mg colchicine a day 20 taking 2.5 mg colchicine a day one blood sample for trough colchicine levels will be taken. response to treatment, colchicine side effects and anthropometric data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* constant colchicine levels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: FMF patients treated with a constant dose of colchicine
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-10-19 (Actual); Primary Completion 2020-07-15 (Estimated); Study Completion 2020-07-15 (Estimated)

PRIMARY OUTCOMES:
colchicine levels | a single measurement under a constant dosage at visit 1 (time=0, recruitment)
  the trough level of colchicine in the serum

CONTACTS AND LOCATIONS:
Overall Officials: merav lidar, prof, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No